CLINICAL TRIAL: NCT01625533
Title: Randomized Study on the Safety and Efficacy of Dual-axis Rotational Versus Standard Coronary Angiography
Brief Title: Safety and Efficacy Study of Dual-axis Rotational Versus Standard Coronary Angiography
Status: Completed | Type: Observational
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Other Study IDs: 20120601
Record Dates: First submitted 2012-06-13; First posted 2012-06-21 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Angiography; Rotational Coronary Angiography; Contrast media; Radiation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- SA group: Patients using SA for the diagnosis of coronary artery disease are assigned to the SA group.
  Interventions: Procedure: Standard Coronary Angiography
- DARCA group: Patients using DARCA for the diagnosis of coronary artery disease are assigned to the DARCA group.
  Interventions: Procedure: Dual-axis Rotational Coronary Angiography

INTERVENTIONS:
Procedure: Standard Coronary Angiography — Using standard coronary angiography (SA) for the diagnosis of coronary artery disease.
  Other Names: Conventional Coronary Angiography
  Groups: SA group
Procedure: Dual-axis Rotational Coronary Angiography — Using dual-axis rotational coronary angiography (DARCA) for the diagnosis of coronary artery disease.
  Other Names: DARA; XPERSWING
  Groups: DARCA group

SUMMARY:
The purpose of this study is to assess the clinical safety and efficacy of dual-axis rotational coronary angiography (DARCA) in the diagnosis of coronary artery disease by directly comparing it to standard coronary angiography (SA).

DETAILED DESCRIPTION:
Dual-axis rotational coronary angiography (DARCA) was developed as an innovative adaptation of rotational angiography (RA), but it requires a longer coronary injection compared to standard coronary angiography (SA). The risk of complications from the contrast agent (such as discomfort, warmth, pain, hypotension and bradycardia) is increased with the use of DARCA. It remains to be evaluated whether this approach is also suitable for coronary angiography, especially using in the patients with complex coronary lesions. Previous studies revealed promising results, but the number of patients included did not provide sufficient statistical power to allow a valid comparison of DARCA with SA. The purpose of this study is to evaluate the feasibility, safety, clinical tolerance, and hemodynamic effect of DARCA in comparison to the well-established SA.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* A clinical indication for diagnostic coronary angiography to evaluate possible CAD

Exclusion Criteria:

* Pregnancy
* Known allergy to iodinated contrast
* Renal insufficiency (>1.5mg/dL)
* Cardiogenic shock
* Acute myocardial infarction within one week
* Prior coronary artery bypass graft treatment
* Prior percutaneous coronary intervention treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing diagnostic coronary angiography at the General Hospital of Chinese People's Armed Police Forces.
Sampling Method: Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2012-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Clinical safety of the patient during coronary angiography(CA) | At time of CA
  The patients were closely observed and questioned regarding discomfort and adverse events during or immediately after CA. The sensation of warmth or pain, including chest pain, is considered as discomfort. Adverse events include arrhythmias, hemodynamic compromise, chest pain described as angina-like pain and any untoward event which jeopardises the patient's life or prolongs the planned hospital stay. If patients experienced bradycardia, only bradycardia with a decrease in heart rate of 20% from the baseline was counted. Hemodynamic compromise was defined as a decrease in systolic blood pressure by > 20 mmHg to < 90 mmHg.

SECONDARY OUTCOMES:
Patient safety determined by contrast and radiation dose | At time of CA
  The contrast usage (ml) and radiation exposure (mGycm2) are recorded from the point of selective catheter engagement in the coronary ostium to the completion of the diagnostic study. The contrast and radiation to perform isocentering are included during DARCA. The contrast and radiation required to engage the coronary ostia, exchange catheters, and perform non-coronary angiography are excluded from the analysis.
Clinical utility of dual-axis rotational coronary angiography(DARCA) | At time of CA
  The clinical utility of DARCA is determined by the number of additional acquisitions required beyond the protocol and the procedure time required for completing CA.The procedure time (sec.) is recorded from the point of selective catheter engagement in the coronary ostium to the completion of the diagnostic study. The time to perform isocentering is included during DARCA. The time required to engage the coronary ostia, exchange catheters, and perform non-coronary angiography is excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Huiliang, M.D., Study Chair — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Jin Zhigeng, M.M., Study Director — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Luo Jianping, M.M., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Yang Shengli, M.D., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Ma Dongxing, M.D., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Liu Ying, M.M., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Han Wei, M.D., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China; Jing Limin, B.S.M., Principal Investigator — Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing 100039, China
Locations (1):
- Division of Cardiology, General Hospital of Chinese People's Armed Police Forces, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Garcia JA, Agostoni P, Green NE, Maddux JT, Chen SY, Messenger JC, Casserly IP, Hansgen A, Wink O, Movassaghi B, Groves BM, Van Den Heuvel P, Verheye S, Van Langenhove G, Vermeersch P, Van den Branden F, Yeghiazarians Y, Michaels AD, Carroll JD. Rotational vs. standard coronary angiography: an image content analysis. Catheter Cardiovasc Interv. 2009 May 1;73(6):753-61. doi: 10.1002/ccd.21918. PMID 19180661
- [Background] Maddux JT, Wink O, Messenger JC, Groves BM, Liao R, Strzelczyk J, Chen SY, Carroll JD. Randomized study of the safety and clinical utility of rotational angiography versus standard angiography in the diagnosis of coronary artery disease. Catheter Cardiovasc Interv. 2004 Jun;62(2):167-74. doi: 10.1002/ccd.20036. PMID 15170705
- [Background] Empen K, Kuon E, Hummel A, Gebauer C, Dorr M, Konemann R, Hoffmann W, Staudt A, Weitmann K, Reffelmann T, Felix SB. Comparison of rotational with conventional coronary angiography. Am Heart J. 2010 Sep;160(3):552-63. doi: 10.1016/j.ahj.2010.06.011. PMID 20826266
- [Background] Gomez-Menchero AE, Diaz JF, Sanchez-Gonzalez C, Cardenal R, Sanghvi AB, Roa-Garrido J, Rodriguez-Lopez JL. Comparison of dual-axis rotational coronary angiography (XPERSWING) versus conventional technique in routine practice. Rev Esp Cardiol (Engl Ed). 2012 May;65(5):434-9. doi: 10.1016/j.recesp.2011.12.014. Epub 2012 Apr 1. English, Spanish. PMID 22465608
- [Background] Grech M, Debono J, Xuereb RG, Fenech A, Grech V. A comparison between dual axis rotational coronary angiography and conventional coronary angiography. Catheter Cardiovasc Interv. 2012 Oct 1;80(4):576-80. doi: 10.1002/ccd.23415. Epub 2012 Jan 12. PMID 22105940
- [Result] Klein AJ, Garcia JA, Hudson PA, Kim MS, Messenger JC, Casserly IP, Wink O, Hattler B, Tsai TT, Chen SY, Hansgen A, Carroll JD. Safety and efficacy of dual-axis rotational coronary angiography vs. standard coronary angiography. Catheter Cardiovasc Interv. 2011 May 1;77(6):820-7. doi: 10.1002/ccd.22804. Epub 2011 Mar 11. PMID 20853352
- [Result] Liu HL, Jin ZG, Yang SL, Luo JP, Ma DX, Liu Y, Han W. Randomized study on the safety and efficacy of dual-axis rotational versus standard coronary angiography in. Chin Med J (Engl). 2012 Mar;125(6):1016-22. PMID 22613524